CLINICAL TRIAL: NCT02903355
Title: Phase 3 Clinical Trial: D-methionine to Reduce Noise-Induced Hearing Loss (NIHL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01345474; NCT01345474 (obsolete NCT alias)
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Noise-induced Hearing Loss
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo contains sorbitol, orange flavor and purified water; is flavor and color matched to D-Met.
  Interventions: Drug: Placebo
- D-methionine, oral liquid suspension (Experimental): D-methionine liquid suspension also contains sorbitol, orange flavor and purified water Intervention: Drug: D-methionine, oral liquid suspension.
  Interventions: Drug: D-methionine

INTERVENTIONS:
Drug: D-methionine — D-methionine, oral liquid suspension
  Arms: D-methionine, oral liquid suspension
Drug: Placebo — Placebo contains sorbitol, orange flavor and purified water; is flavor and color matched to D-Met.
  Arms: Placebo

SUMMARY:
This prospective study is a randomized, double-blind, placebo-controlled Phase 3 clinical trial of oral D-methionine (D-met) to reduce noise-induced hearing loss (NIHL) and tinnitus. The goal of the study is to develop a safe, oral pharmacological agent to augment physical hearing protectors for noise exposures that exceed the protective capabilities of ear plugs and/or muffs. The study population is a cohort of Drill Sergeant (DS) instructor trainees during and 22 days after their 11 day weapons training. The primary objective of this study is to determine the efficacy of D-met in preventing NIHL or reducing tinnitus secondary to a minimum of 500 rounds of M-16 weapons training occurring over an 11 day period.

DETAILED DESCRIPTION:
Hearing loss can render a soldier less able to detect and identify the enemy, less able to understand commands, particularly in background noise typical on the battlefield, and may permanently reduce quality of life. In some cases, hearing loss may preclude redeployment or result in less optimal job assignment. Currently, no FDA approved pharmacological prevention exists for noise-induced hearing loss (NIHL). We have documented in animal studies that administration of D-methionine (D-met) can reduce or prevent NIHL. We now need to determine if it has similar efficacy in humans. Although we have not yet tested D-met on protection from noise-induced tinnitus in animals, this clinical trial would provide us the opportunity to also test for protection from noise induced tinnitus simultaneously.

Objective Hypotheses:

Primary Hypothesis: Administration of oral D-methionine prior to, during and 4 days post-weapons training will reduce or prevent permanent noise-induced hearing loss.

Secondary Hypothesis: Administration of oral D-methionine prior to, during and 4 days post-weapons training will reduce or prevent noise-induced tinnitus.

Specific Aims:

To determine whether administering oral D-met can prevent permanent NIHL after weapons training. This aim will be addressed by comparing the results of D-met versus placebo administration starting 3 days prior to, during the 11 day period of weapons training (Monday-Friday for first week, Monday-Thursday for second week), and 4 days after for a total of 18 days. Pure tone hearing thresholds will be assessed before and 22 days after completion of weapons training (ie; 18 days after the last day of study drug/placebo administration).

To determine whether administering oral D-met can prevent tinnitus after weapons training. This aim will be addressed by comparing the results of D-met versus placebo administration starting 3 days prior to, during the 11 day period of weapons training (Monday-Friday for first week, Monday-Thursday for second week), and 4 days after for a total of 18 days. Tinnitus questionnaires will be assessed before and 22 days after completion of weapons training (ie; 18 days after the last day of study drug/placebo administration).

To monitor for any potential side effects of D-met in human subjects. This aim will be accomplished by subject query on each day study drug is dispensed (twice daily) and at final study visit, routing of any adverse event reports to study medical personnel, statisticians and to the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion criteria:

Male or female 21 to 45 years of age Negative pregnancy test at enrollment and prior to taking study drug Willing to use an effective method of birth control during the study (Both male and female participants should avoid pregnancy during study) Pure tone air conduction threshold average at 0.5, 1 and 2 kHz of no greater than 40 dB HL bilaterally with no air bone gaps greater than 10 dB and normal otoscopy and tympanometry screens Willing to refrain from using supplements containing or derived from protein while participating in this study Ability to comply with all study requirements

Exclusion criteria:

History of allergic or idiosyncratic reaction to methionine, amino acid mixtures, nutritional supplements, egg white, or other proteins or food additives Vegetarian (Individual excludes meat and fish from their diet) History of chronic balance disorders Abnormal otoscopic findings, otologic surgery, autoimmune inner ear disease, significant air-bone gaps, abnormal tympanograms or other indication of middle-ear abnormality, history of fluctuant hearing or asymmetric hearing worse than 25 dB at any frequency in either ear, perilymphatic fistula, tumor of the auditory system, or other CNS disorder that is likely to affect hearing Treatment with intravenous (IV) antibiotics within the past 6 months Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of any drug Treatment for alcohol or substance abuse within past 6 months Women of childbearing age who are not using effective contraceptive methods and who may become pregnant during the course of the study Women who are pregnant or breastfeeding. National Guardsmen History of psychotic schizophrenia Exposure within the previous 6 months to systemic ototoxic substances including aminoglycosides or vancomycin Body weight exceeding 225 pounds Renal impairment measured as eGFR < 50 on screening creatinine clearance blood draw.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Campbell, PhD, Principal Investigator — MetArmor, Inc.; CPT William Grimes, MD, Study Director — United States Department of Defense, US Army Ft. Jackson, South Carolina
Locations (1):
- Moncrief Army Community Hospital, Fort Jackson, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Started | 186 | 165
Completed | 142 | 124
Not Completed | 44 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension | Total
Number analyzed (Participants) | 142 | 124 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 142 | 124 | 266
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.34 (4.01) | 31.01 (4.35) | 30.65 (4.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 108 | 97 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Hispanic | 32 | 29 | 61
  Asian or Native Hawaiian or Pacific Islander | 4 | 4 | 8
  Black or African American | 18 | 17 | 35
  White | 84 | 73 | 157
  More than on race | 1 | 0 | 1
  Unknown or not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 142 | 124 | 266

OUTCOME MEASURES:

1. Primary Outcome: ASHA Shift Ear (Left)
Description: An increase of at least 20 dB at any one frequency,
  An increase of at least 10 dB at any two consecutive frequencies, or
  Loss of response at 3 consecutive frequencies where responses were obtained at baseline.
Time Frame: Change from baseline to day 29-36 after initial administration of study drug (Day 15-22 after cessation of weapons training).
Population: 5 and 3 participants in the placebo and D-methionine arms, respectively, failed a final tympanogram screen in the left ear to rule out middle ear pathology as a cause of the hearing loss and were excluded from the analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 137 | 121
Participants | 12 | 9
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .4385, Fisher Exact

2. Primary Outcome: ASHA Shift Ear (Right)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 3 and 4 participants in the placebo and D-methionine arms, respectively, failed a final tympanogram screen in the right ear to rule out middle ear pathology as a cause of the hearing loss and were excluded from the analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 139 | 120
Participants | 12 | 10
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .5562, Fisher Exact

3. Primary Outcome: ASHA Shift Ear (Either)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 7 and 7 participants in the placebo and D-methionine arms, respectively, failed a final tympanogram screen in either ear to rule out middle ear pathology as a cause of the hearing loss and were excluded from the analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 135 | 117
Participants | 21 | 18
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .5441, Fisher Exact

4. Primary Outcome: ASHA Shift Ear (Both)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 135 | 117
Participants | 3 | 1
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .3666, Fisher Exact

5. Primary Outcome: ASHA Shift Ear (Trigger Hand)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 3 and 4 participants in the placebo and D-methionine arms, respectively, failed a final tympanogram screen in the trigger hand ear to rule out middle ear pathology as a cause of the hearing loss and were excluded from the analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 139 | 120
Participants | 11 | 8
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .4446, Fisher Exact

6. Primary Outcome: ASHA Shift Ear (Non-Trigger Hand)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 5 and 3 participants in the placebo and D-methionine arms, respectively, failed a final tympanogram screen in the non-trigger hand ear to rule out middle ear pathology as a cause of the hearing loss and were excluded from the analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 137 | 121
Participants | 13 | 11
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .5431, Fisher Exact

7. Secondary Outcome: DOEHRSHC Shift
Description: Greater than or equal to 10 dB change for the average of 2k, 3k, and 4k in either ear. This is a binary outcome measure based on meeting this definition.
Time Frame: as for outcome 1
Population: 0 and 1 participants in the placebo and D-methionine arms, respectively, failed a final tympanogram screen in both ears to rule out middle ear pathology as a cause of the hearing loss and were excluded from the analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 142 | 123
Participants | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .7409, Fisher Exact

8. Secondary Outcome: EWS STS Shift
Description: Greater than or equal to 15 dB change (deficit) in any of the following frequencies in either ear (1k or 2k or 3k or 4k). This is a binary outcome measure based on meeting this definition.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 142 | 123
Participants | 11 | 5
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .1597, Fisher Exact

9. Secondary Outcome: Total THI Score Change
Description: Tinnitus Handicap Inventory. Tinnitus handicap inventory designed to evaluate the difficulties experienced as a result of hearing loss. Score ranges from 0 to 100 with 0 indicating no handicap, and 100 indicating catastrophic handicap. The THI score was to compare pre and post treatment effects of hearing loss.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 142 | 124
units on a scale | .169 (5.3022) | -.1452 (3.2876)
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .2784, t-test, 1 sided

10. Secondary Outcome: Significant Change in Tinnitus
Description: An increase of at least 5 points in the Tinnitus Handicap Inventory (THI), AND an increase in one severity grade category (Categories listed below). Tinnitus handicap inventory is designed to evaluate the difficulties experienced as a result of hearing loss. Score ranges from 0 to 100, with 0 indicating no handicap, and 100 indicating catastrophic handicap. The THI score was to compare pre and post treatment effects of hearing loss.
  0-16: Slight or no handicap (Grade 1) 18-36: Mild handicap (Grade 2) 38-56: Moderate handicap (Grade 3) 58-76: Severe handicap (Grade 4) 78-100: Catastrophic handicap (Grade 5)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
Number analyzed (Participants) | 142 | 124
Participants | 4 | 1
Statistical Analysis 1: Comparison: Placebo vs D-methionine, Oral Liquid Suspension; Test type: Superiority; p = .2303, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events monitored from first dose to day 36.
Description: The at-risk numbers presented are for those subjects that took at least one dose (D-Met or placebo). If they did not take a dose, even if they started the study, they were not considered at risk for an adverse event.
Arm/Group | Placebo | D-methionine, Oral Liquid Suspension
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/157
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/157
Other Adverse Events (participants affected / at risk) | 93/159 | 120/157
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | D-methionine, Oral Liquid Suspension (N=157)
Abdominal Pain/Cramps (Gastrointestinal disorders) | 6 | 9
Body Odor (Product Issues) | 3 | 35
Diarrhea (Gastrointestinal disorders) | 12 | 18
Flatulence (Product Issues) | 56 | 52
Headache (Nervous system disorders) | 9 | 9
Nausea/ Vomiting (Gastrointestinal disorders) | 10 | 27
Urine Odor (Product Issues) | 7 | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT02903355/Prot_SAP_000.pdf